CLINICAL TRIAL: NCT01876316
Title: A Randomized, Double-blind, Placebo-controlled, Two-way Crossover Trial to Compare Moxifloxacin Induced QT Interval Prolongation in Japanese and Korean Healthy Subjects
Brief Title: The Effect of Ethnic on Moxifloxacin Induced QT Interval Prolongation in Korean and Japanese Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jae-Gook Shin, Department of Pharmacology and Pharmacogenomics Research Center, Inje University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 12-166
Record Dates: First submitted 2013-06-09; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Moxifloxacin; QT interval prolongation; Korean; Japanese
MeSH Terms: interventions — Moxifloxacin; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Active Comparator): single oral administration of 400mg of moxifloxacin
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): single oral administration of 400mg of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — single oral administration of 400mg of moxifloxacin
  Other Names: Avelox
  Arms: Moxifloxacin
Drug: Placebo — single oral administration of 400mg of placebo
  Other Names: Lactose
  Arms: Placebo

SUMMARY:
The Effect of Ethnic on Moxifloxacin Induced QT Interval Prolongation in Korean and Japanese Healthy Subjects

DETAILED DESCRIPTION:
The purpose of this study is to explore the ethnic and gender difference in the Moxifloxacin induced QT interval prolongation between Japanese and Korean subjects.

ELIGIBILITY:
Inclusion Criteria:

- 1) Subjects in Japan and Korea deemed healthy as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, or clinical laboratory determinations.

2) Body Mass Index (BMI) of 17.6 to 26.4 kg/m2, BMI = weight (kg)/ [height (m)]2.

Exclusion Criteria:

* 1) Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population.

  2) Any of the following on 12-lead ECG prior to study drug administration, confirmed by repeat.
* Heart rate ≤ 45 bpmmsec or Heart rate ≥ 100 bpmmsec
* PR ≥ 210 msec
* QRS ≥ 120 msec
* QT ≥ 500 msec
* QTcF: male ≥ 450 msec, female ≥470msec
* Iincomplete right bundle branch block
* Marked Sinus Arrhythmia
* Wondering pacemaker
* Atrial rhythm

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
double delta QTcF | up to 24 hours
  12 point of ECG measurements according to the interventions

SECONDARY OUTCOMES:
double delta QTcI, double delta QTcSS | up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Gook Shin, MD, PhD, Principal Investigator — Inje University

REFERENCES:
- [Derived] Choi HK, Jung JA, Fujita T, Amano H, Ghim JL, Lee DH, Tabata K, Song ID, Maeda M, Kumagai Y, Mendzelevski B, Shin JG. Population Pharmacokinetic-Pharmacodynamic Analysis to Compare the Effect of Moxifloxacin on QT Interval Prolongation Between Healthy Korean and Japanese Subjects. Clin Ther. 2016 Dec;38(12):2610-2621. doi: 10.1016/j.clinthera.2016.10.011. PMID 28003052